CLINICAL TRIAL: NCT02776462
Title: Use of Eye Movement Tracking to Detect Oculomotor Abnormality in Traumatic Brain Injury Patients
Acronym: DETECT
Status: Completed | Type: Observational
Sponsor: Oculogica, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: DETECT TBI001
Record Dates: First submitted 2016-05-16; First posted 2016-05-18 (Estimated); Last update posted 2018-09-07 (Actual); Status verified 2018-09

CONDITIONS: Brain Concussion; Cerebral Concussion; Concussion, Intermediate; Concussion, Mild; Concussion, Severe; Trauma, Nervous System; Craniocerebral Trauma; Brain Injuries
Keywords: Eye Tracking; Concussion; Outcome Measures
MeSH Terms: conditions — Brain Concussion; Trauma, Nervous System; Craniocerebral Trauma; Brain Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Potential Traumatic Brain Injury: This group will consist of people admitted to the ER, Trauma Bay, or Neurosurgery for potential traumatic brain injury.
  Interventions: Device: EyeBox CNS

INTERVENTIONS:
Device: EyeBox CNS

SUMMARY:
The purpose of this study is to determine the sensitivity and specificity of an aid in assessment of concussion based on eye-tracking, in comparison to a clinical reference standard appropriate for the Emergency Department (ED) or concussion clinic.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent.
* Be between the ages of 4 and 67 years old.
* Have a diagnosis of traumatic brain injury with a potential for concussion.
* Subjects must have baseline vision correctable to within 20/500 bilaterally.
* Subjects must have intact ocular motility.
* Subjects must have ability to provide a complete ophthalmologic, medical and neurologic history as well as medications/drugs/alcohol consumed within the 24 hours prior.

Exclusion Criteria:

* ER visit has been more than 2 weeks since the injury which may have caused the concussion.
* Have received penetrating trauma or have a head CT demonstrating evidence of acute brain injury (subdural, epidural or intraparenchymal hemorrhage, edema/mass effect per attending radiologist read).
* Suffering burns, anoxic injury or multiple/extensive injuries resulting in any medical, surgical or hemodynamic instability.
* Blind (no light perception), are missing eyes, do not open eyes.
* It is pertinent that subjects be able to detect light and have both eyes in order for the eye tracking data to be effective and significant.
* Previous history of: ocular motility dysfunction or extensive prior eye surgery.
* Any physical or mental injury or baseline disability rendering task completion difficult.
* Obvious intoxication or blood alcohol level greater than 0.2.

Ages: 5 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants will include all patients evaluated for potential traumatic brain injury presenting to the Emergency Department or concussion clinic.
Sampling Method: Probability Sample
Enrollment: 321 (Actual)
Dates: Start 2016-06; Primary Completion 2017-11-16 (Actual); Study Completion 2018-06-19 (Actual)

PRIMARY OUTCOMES:
A change in metrics of eye movement that enable positive concussion detection using BOX Score. | Immediately after eye tracking, within 2 weeks of injury
  A True Positive rate for identifying Concussion as compared to a Clinical Reference standard.

SECONDARY OUTCOMES:
Change in Cognitive Function and Symptom Severity during Recovery as Measured with a Clinical Reference Standard for Concussion. | Immediately before eye tracking, between 1 week and 109 weeks post injury

CONTACTS AND LOCATIONS:
Overall Officials: Uzma Samadani, M.D., Ph.D., Study Chair — Hennepin County Medical Center, Minneapolis
Locations (2):
- United States (2):
  - SkyRidge Medical Center, Lone Tree, Colorado
  - Beaver Dam Community Hospital, Beaver Dam, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Samadani U. A new tool for monitoring brain function: eye tracking goes beyond assessing attention to measuring central nervous system physiology. Neural Regen Res. 2015 Aug;10(8):1231-3. doi: 10.4103/1673-5374.162752. No abstract available. PMID 26487847
- [Background] Samadani U, Ritlop R, Reyes M, Nehrbass E, Li M, Lamm E, Schneider J, Shimunov D, Sava M, Kolecki R, Burris P, Altomare L, Mehmood T, Smith T, Huang JH, McStay C, Todd SR, Qian M, Kondziolka D, Wall S, Huang P. Eye tracking detects disconjugate eye movements associated with structural traumatic brain injury and concussion. J Neurotrauma. 2015 Apr 15;32(8):548-56. doi: 10.1089/neu.2014.3687. Epub 2015 Feb 6. PMID 25582436
- [Background] Samadani U, Farooq S, Ritlop R, Warren F, Reyes M, Lamm E, Alex A, Nehrbass E, Kolecki R, Jureller M, Schneider J, Chen A, Shi C, Mendhiratta N, Huang JH, Qian M, Kwak R, Mikheev A, Rusinek H, George A, Fergus R, Kondziolka D, Huang PP, Smith RT. Detection of third and sixth cranial nerve palsies with a novel method for eye tracking while watching a short film clip. J Neurosurg. 2015 Mar;122(3):707-20. doi: 10.3171/2014.10.JNS14762. Epub 2014 Dec 12. PMID 25495739